CLINICAL TRIAL: NCT07408089
Title: An Open-Label, Multicenter, First-in-Human, Phase 1 Study of BBI-940 in Advanced or Metastatic Breast Cancer: Kinesin Oral Molecular Degrader for Oncology (KOMODO-1)
Brief Title: Study of the Kinesin Oral Molecular Degrader BBI-940 in Subjects With Advanced or Metastatic Breast Cancer
Acronym: KOMODO-1
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boundless Bio (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BBI-940-101
Record Dates: First submitted 2026-01-22; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Advanced Breast Cancer
Keywords: Breast Cancer; Metastatic Breast Cancer; Advanced Breast Cancer; Phase 1; First in Human; BBI-940; Fulvestrant
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Intervention Model Description: BBI-940 single agent dose escalation and expansion, and BBI-940 dose expansion (at multiple potential dose levels) in combination with fulvestrant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Parts 1A, 1B. BBI-940 Monotherapy Escalation (Experimental): Participants receive BBI-940 given alone in multiple sequential dose escalation cohorts. BBI-940 is given orally in repeated 28-day cycles.
  Interventions: Drug: BBI-940
- Part 2A. BBI-940 in Combination with Fulvestrant (ER+/HER2- Breast Cancer without an ESR1 Mutation) (Experimental): Participants receive BBI-940 in combination with fulvestrant. BBI-940 is given orally in repeated 28-day cycles at one of multiple potential dose levels.
  Interventions: Drug: BBI-940; Drug: Fulvestrant
- Part 2B. BBI-940 Monotherapy Expansion (ER+/HER2- Breast Cancer with FGFR1 Amplification) (Experimental): Participants receive BBI-940 given alone at the recommended dose for expansion (RDE). BBI-940 is given orally in repeated 28-day cycles.
  Interventions: Drug: BBI-940
- Part 2C. BBI-940 Monotherapy Expansion (TNBC-LAR) (Experimental): Participants receive BBI-940 given alone at the recommended dose for expansion (RDE). BBI-940 is given orally in repeated 28-day cycles.
  Interventions: Drug: BBI-940

INTERVENTIONS:
Drug: BBI-940 — Oral small molecule degrader targeting Kinesin.
Drug: Fulvestrant — Selective estrogen receptor degrader administered intramuscularly.
  Arms: Part 2A. BBI-940 in Combination with Fulvestrant (ER+/HER2- Breast Cancer without an ESR1 Mutation)

SUMMARY:
This is a first-in-human, open-label, Phase 1 study evaluating BBI-940, an investigational kinesin oral molecular degrader, administered as monotherapy or in combination with fulvestrant in adults with advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
The study consists of two parts: Part 1 (dose escalation) and Part 2 (dose expansion).

Part 1 is a dose-escalation phase designed to evaluate the safety and tolerability of BBI-940 and to determine the recommended dose for expansion (RDE). Participants may have estrogen receptor-positive, HER2-negative (ER+/HER2-) breast cancer or triple-negative breast cancer of the luminal androgen receptor subtype (TNBC-LAR).

Part 2 is a dose-expansion phase designed to further evaluate BBI-940 at the selected RDE in defined participant populations.

Part 2A evaluates BBI-940 in combination with fulvestrant, including multiple dose cohorts to evaluate the safety of the combination regimen and to determine the combination RDE in participants with ER+/HER2- breast cancer without an ESR1 mutation.

Part 2B evaluates BBI-940 monotherapy at the RDE in participants with ER+/HER2- breast cancer with FGFR1 amplification.

Part 2C evaluates BBI-940 monotherapy at the RDE in participants with TNBC-LAR.

Across all parts of the study, treatment is administered in repeated 28-day cycles, and participants undergo protocol-specified safety assessments.

ELIGIBILITY:
Key Inclusion Criteria

* Adults with locally advanced or metastatic breast cancer, including estrogen receptor-positive/human epidermal growth factor receptor 2-negative (ER+/HER2-) disease or triple-negative breast cancer with luminal androgen receptor subtype (TNBC-LAR; androgen receptor expression ≥10% by immunohistochemistry), as applicable by study part.
* Prior treatment with standard therapies known to provide clinical benefit, appropriate for disease subtype and study part, including endocrine therapy with CDK4/6 inhibition for ER+/HER2- disease.
* Measurable disease per RECIST v1.1, except for participants enrolled in Part 1A.
* Molecular eligibility as applicable by study part, including absence of an ESR1 mutation (Part 2A) or presence of FGFR1 amplification (Part 2B), based on prior local testing.
* Availability of archival or newly obtained formalin-fixed, paraffin-embedded (FFPE) tumor tissue suitable for protocol-specified biomarker analyses.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Adequate hematologic, hepatic, renal, and coagulation function per protocol-defined laboratory criteria.
* Estimated life expectancy of at least 12 weeks.
* Ability to swallow oral medication and provide written informed consent.

Key Exclusion Criteria

* Prior exposure to an inhibitor or degrader of Kinesin.
* Known hypersensitivity to study intervention(s) or excipients.
* Receipt of recent anticancer therapy within protocol-defined washout periods.
* Other active malignancy likely to interfere with study assessment.
* Baseline QTcF >470 msec or congenital long QT syndrome.
* Clinically significant pulmonary embolism within 6 weeks prior to first dose.
* Major surgery within 4 weeks or minor surgery within 2 weeks prior to first dose.
* Active infection requiring systemic therapy within 2 weeks prior to first dose.
* Pregnant or breastfeeding, or planning conception or gamete donation during the study or required post-treatment period.
* Prior solid organ transplant or allogeneic stem cell transplant with protocol-defined exceptions.
* Failure to recover to CTCAE Grade ≤1 (or baseline) from prior anticancer therapy, with protocol-specified exceptions.
* Any serious or uncontrolled medical, laboratory, or psychiatric condition that could compromise safety or study integrity.
* Other exclusion criteria as specified in the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities (DLTs) in each BBI-940 monotherapy dose escalation cohort. | First 28 days of study treatment (through end of Cycle 1).
  DLTs will be assessed during the first 28 days of study treatment (Cycle 1) to establish the maximum tolerated dose (MTD) and the recommended dose for expansion (RDE) of BBI-940 as monotherapy.
Incidence of treatment emergent adverse events (TEAEs) in each dose group and overall as assessed by CTCAE version 5.0. | First dose of study treatment through 30 days after the last dose of study treatment.
  Incidence of treatment emergent adverse events (TEAEs) will be assessed by maximum severity and maximum causality.
Incidence of study treatment discontinuation and/or interruption by dose group and overall. | First dose of study treatment through 30 days after the last dose of study treatment.
  The incidence of study treatment discontinuation and/or interruption will be assessed.

SECONDARY OUTCOMES:
Objective response rate (ORR) per RECIST Version 1.1 by dose group and overall. | From first dose of study treatment until disease progression per RECIST 1.1, death, withdrawal, loss to follow-up, or study completion; tumor assessments every 8 weeks (±7 days); assessed up to approximately 3 years.
  Objective response rate (ORR) will be summarized by dose group and overall, based on the number of participants achieving a best response of partial response or complete response.
Progression Free Survivial (PFS) per RECIST Version 1.1 by dose group and overall. | From first dose of study treatment until first documented disease progression per RECIST 1.1 or death from any cause, whichever occurs first; tumor assessments every 8 weeks (±7 days); assessed up to approximately 3 years.
  Progression-free survival is defined as the time from first dose of study treatment to the first documented disease progression per RECIST Version 1.1 or death from any cause, whichever occurs first.
Time of maximum plasma concentration (Tmax) of BBI-940. | From 0 hours through up to 24 hours after BBI-940 dosing.
  Time of maximum plasma concentration (Tmax) of BBI-940 will be determined.
Maximum observed plasma concentration (Cmax) of BBI-940. | From 0 hours through up to 24 hours after BBI-940 dosing.
  Maximum observed plasma concentration (Cmax) of BBI-940 will be determined.
Minimum observed plasma concentration (Ctrough) of BBI-940. | From 0 hours through up to 24 hours after BBI-940 dosing.
  Minimum observed plasma concentration (Ctrough) of BBI-940 will be determined.
Area under the plasma concentration-time curve (AUC) of BBI-940. | From 0 hours through up to 24 hours after BBI-940 dosing.
  Area under the plasma concentration-time curve (AUC) of BBI-940 will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Doebele, MD, PhD, Study Director — Boundless Bio

IPD SHARING:
Plan to Share IPD: No